CLINICAL TRIAL: NCT00143793
Title: Mannheim NT-proBNP Study (MANPRO) Evaluating NT-proBNP and New Biomarkers in Patients Suffering From Dyspnea and/or Peripheral Edema for the Differential Diagnosis of Congestive Heart Failure
Brief Title: NT-proBNP and New Biomarkers in Patients With Dyspnea and/or Peripheral Edema
Acronym: MANPRO
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Michael Behnes, Dr. med., Universitätsmedizin Mannheim
Other Study IDs: 80/05
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Dyspnea; Peripheral Edema
Keywords: natruretic peptides; NT-proBNP; new biomarkers; congestive heart failure; atrial fibrillation; acute myocardial infarction; lung embolism
MeSH Terms: conditions — Dyspnea; Heart Failure; Atrial Fibrillation; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of this study are to:

* Evaluate the sensitivity and specificity of NT-proBNP (N-terminal prohormone brain natriuretic peptide) and new biomarker measurements for the diagnosis of heart failure in patients with acute dyspnea and/or edema.
* Determine the exact biomarker cut-off point(s) for the differentiation of healthy persons, patients with heart failure and patients with dyspnea of other origin.
* Evaluate treatment costs in patients with dyspnea under special consideration of NT-proBNP measurement.

DETAILED DESCRIPTION:
Primary endpoint:

* Sensitivity and specificity of biomarker measurements for discrimination of heart failure from dyspnea of other origin.

Secondary endpoints:

* Determination of Cut-off(s)
* Discrimination of cardiac and non-cardiac diseases causing to dyspnea or peripheral edema
* Determination of treatment costs of the initial hospital stay
* Evaluation of resource savings when implementing NT-proBNP for determination of diagnosis.
* Time to diagnosis.
* Hospitalization rate /Intensive care treatment rate between day 1 and 28
* Duration of initial hospital stay
* 30-day re-hospitalization rate
* 30 day mortality rate and adverse event rate
* 1 and 5 year mortality rates
* 1 and 5 year rehospitalization rates

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years
* Dyspnea or/and peripheral edema
* Informed consent

Exclusion Criteria:

* Renal insufficiency with creatinine > 2.8mg/dl
* Anemia (hemoglobin < 8.0mg/dl)
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from dyspnea and peripheral edema
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2005-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martina Brueckmann, MD, Study Chair — First Department of Medicine, University Medical Centre Mannheim; Martin Borggrefe, MD, Study Chair — First Department of Medicine, University Medical Centre Mannheim; Michael Neumaier, MD, Principal Investigator — Institute of Clinical Chemistry, University Medical Centre Mannheim; Parviz Ahmad-Nejad, MD, Study Chair — Institute of Clinical Chemistry, University Medical Centre Mannheim; Michael Behnes, MD, Principal Investigator — First Department of Medicine, University Medical Centre Mannheim; Ursula Hoffmann, MD, Study Chair — First Department of Medicine, University Medical Centre Mannheim
Locations (1):
- Medical Faculty Mannheim, University of Heidelberg, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Hoffmann U, Espeter F, Weiss C, Ahmad-Nejad P, Lang S, Brueckmann M, Akin I, Neumaier M, Borggrefe M, Behnes M. Ischemic biomarker heart-type fatty acid binding protein (hFABP) in acute heart failure - diagnostic and prognostic insights compared to NT-proBNP and troponin I. BMC Cardiovasc Disord. 2015 Jun 14;15:50. doi: 10.1186/s12872-015-0026-0. PMID 26072112
- [Derived] Behnes M, Brueckmann M, Lang S, Weiss C, Ahmad-Nejad P, Neumaier M, Borggrefe M, Hoffmann U. Connective tissue growth factor (CTGF/CCN2): diagnostic and prognostic value in acute heart failure. Clin Res Cardiol. 2014 Feb;103(2):107-16. doi: 10.1007/s00392-013-0626-6. Epub 2013 Oct 22. PMID 24146089
- [Derived] Behnes M, Brueckmann M, Lang S, Espeter F, Weiss C, Neumaier M, Ahmad-Nejad P, Borggrefe M, Hoffmann U. Diagnostic and prognostic value of osteopontin in patients with acute congestive heart failure. Eur J Heart Fail. 2013 Dec;15(12):1390-400. doi: 10.1093/eurjhf/hft112. Epub 2013 Jul 12. PMID 23851388